CLINICAL TRIAL: NCT00133081
Title: Study to Improve the Treatment of Epilepsy (SITE). A Randomized Study Comparing Adjustment of Treatment to Reduce Side Effects of Antiepileptic Drugs With Continuing Treatment Unchanged
Brief Title: Study to Improve the Treatment of Epilepsy (SITE)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SITE
Record Dates: First submitted 2005-08-17; First posted 2005-08-22 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2004-03

CONDITIONS: Epilepsy
Keywords: epilepsy; antiepileptic drugs; side effects; quality of life
MeSH Terms: conditions — Epilepsy

INTERVENTIONS:
Drug: All registered antiepileptic drugs

SUMMARY:
The purpose of this study is to assess whether changing antiepileptic medication can reduce side effects and improve the quality of life in patients with epileptic seizures that are well controlled with antiepileptic drugs.

DETAILED DESCRIPTION:
Background. The aim of the treatment with antiepileptic drugs (AEDs) is to achieve seizure freedom without causing side effects. Assessment of side effects is difficult. They may start insidiously, the patient may not associate certain complaints with the use of AEDs, or the treating physician does not take enough time to discuss this topic during the limited time of a visit in the outpatient department. We know from clinical trials that side effects occur in a substantial group of patients. We do not know whether we deal with this possible complication in an adequate way in clinical practice.

Study objective. To study whether adjustment of medication will reduce the occurrence of side effects and improve quality of life.

Study design. A randomised clinical trial comparing adjustment of treatment in case of relevant side effects to continuing treatment unchanged. Relevant side effects are defined as at least one moderate or serious problem scored on a questionnaire to assess complaints in people with epilepsy.

Patients who do not report relevant side effects will be followed for 13 months (arm A) in which two visits are scheduled, after 7 and 13 months respectively.

The patients who do report relevant side effects will be randomised to either discussion of the questionnaire results and adjustment of treatment if appropriate (arm B) or to ignore the results of the questionnaire and continue treatment unchanged (arm C). Investigations will be repeated in both groups after 7 and 13 months after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Treatment: antiepileptic drugs for epilepsy
* No change in medication during last 6 months
* No obvious clinical reason to change medication immediately

Exclusion Criteria:

* Concurrent disease or disorder that might interfere with the conduct of the study
* Inability to comply to the protocol
* Impaired intellectual functioning, leading to inability to comply to the protocol and complete the necessary questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255
Dates: Start 2002-10; Study Completion 2006-08

PRIMARY OUTCOMES:
Complaints (questionnaire) at 7 and 13 months

SECONDARY OUTCOMES:
Quality of Life (Qolie-10) at 7 and 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Cees A van Donselaar, MD PhD, Study Director — UMC Utrecht; Sabine G Uijl, MSc, Principal Investigator — UMC Utrecht; Albert P Aldenkamp, PhD, Principal Investigator — AZM Maastricht; Cuno SP Uiterwaal, PhD, Principal Investigator — UMC Utrecht
Locations (6):
- Netherlands (6):
  - AZM, Maastricht, Limburg
  - Catharina Hospital, Eindhoven, North Brabant
  - Hospital Gooi-Noord, Blaricum, North Holland
  - MCRZ, Rotterdam, South Holland
  - MC Haaglanden, The Hague, South Holland
  - Oosterschelde Hospital, Goes, Zeeland